CLINICAL TRIAL: NCT04077632
Title: Effects of Transcranial Direct Current Stimulation on Heart Rate Variability in Chronic Low Back Pain Patients: a Randomized Controlled Trial
Brief Title: Effects of tDCS on Heart Rate Variability in Chronic Low Back Pain
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidade Federal do Piauí (Other)
Responsible Party: Principal Investigator, Fuad Ahmad Hazime, Clinical Professor - Physical Therapy Department, Universidade Federal do Piauí
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: tDCS and HRV
Record Dates: First submitted 2019-08-28; First posted 2019-09-04 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Chronic Low-back Pain
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS (anodal) (Experimental): Real transcranial direct current stimulation tDCS: 20 minutes, 2mA, primary motor cortex anode (contralateral to the lesion) and supraorbital cathode (ipsilateral to the lesion).
  Interventions: Device: Transcranial direct current stimulation
- tDCS (sham) (Sham Comparator): Sham transcranial direct current stimulation tDCS: 20 minutes (30 seconds ON), 2mA, primary motor cortex anode (contralateral to the lesion) and supraorbital cathode (ipsilateral to the lesion).
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — tDCS: 20 minutes, 2mA, primary motor cortex anode (contralateral to the lesion) and supraorbital cathode (ipsilateral to the lesion).Technique based on the application of weak, direct electrical current to the brain through relatively large electrodes that are placed over the scalp, in which anodal and cathodal stimulation increases and decreases cortical excitability, respectively.

SUMMARY:
Chronic low back (CLBP) pain is an important public health and socioeconomic problem worldwide and, despite the volume of research in the area, it remains a difficult condition to treat. There are some evidences that altered heart rate variability (HRV) parameters are associated with different clinical disorders, such as chronic low back pain. For instances, diminished parasympathetic activity has been explored as a potential therapeutic target. Considering the dynamic interaction between brain and heart, neuromodulatory strategies targeting this relationship could exert a positive influence on cardiac autonomic system and pain modulation systems.

Transcranial direct current (tDCS) stimulation is a noninvasive neuromodulation technique that has been presenting recent advances in the treatment of chronic pain. However, tDCS application focusing on brain-heart interaction has not been extensively explored, especially on chronic pain conditions.

This study aims to investigate the effects of tDCS on HRV in chronic low back pain patients. Sixty patients will be randomized into two distinct groups to receive either tDCS (anodal) or tDCS (sham) in a single session protocol. The primary clinical outcome (HRV parameter) will be collected before, during and post-tDCS. The data will be collected by a blind examiner to the treatment allocation.

ELIGIBILITY:
Inclusion Criteria:

* Complaining of back pain for more than three months.
* Presence of a chronic pain measurable with the number rating scale (NRS 0-10) not less than 4 during a 1 week daily NRS monitoring.
* Seeking care for low back pain.

Exclusion Criteria:

* Previous surgery on the spine
* Spondylolisthesis
* Previous treatment with tDCS
* Disc herniation with nerve compression Neurological
* Psychiatric
* Rheumatologic diseases
* Impaired sensibility
* Use of pacemakers or other implanted devices
* Pregnancy
* Cardiovascular diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
HRV frequency-domain measures | After 13 minutes of tDCS
  Frequency domain analysis is conducted to evaluate two components: high frequency (HF) (0.14 and 0.40 Hz), related to the parasympathetic nervous system, and low frequency (LF) (0.004 and 0.15 Hz), related to the sympathetic and parasympathetic nervous system, with predominance of the sympathetic component
HRV time-domain measures | After 13 minutes of tDCS
  Time domain analysis is related to global autonomic modulation and is conducted to evaluate differences between RR normal intervals (NN), defined as the temporal distance between consecutive "normal" beats (sinoatrial depolarizations) between the R peaks of the QRS complex, and their measurements including standard deviation of NN intervals (SDNN), standard deviation of mean RR intervals (SDANN), root mean square differences of successive RR intervals (RMSSD), and the percentage of normal RR intervals that differ by 50 ms (pNN50).

SECONDARY OUTCOMES:
HRV frequency-domain measures | After 20 minutes of tDCS
  Frequency domain analysis is conducted to evaluate two components: high frequency (HF) (0.14 and 0.40 Hz), related to the parasympathetic nervous system, and low frequency (LF) (0.004 and 0.15 Hz), related to the sympathetic and parasympathetic nervous system, with predominance of the sympathetic component
HRV time-domain measures | After 20 minutes of tDCS
  Time domain analysis is related to global autonomic modulation and is conducted to evaluate differences between RR normal intervals (NN), defined as the temporal distance between consecutive "normal" beats (sinoatrial depolarizations) between the R peaks of the QRS complex, and their measurements including standard deviation of NN intervals (SDNN), standard deviation of mean RR intervals (SDANN), root mean square differences of successive RR intervals (RMSSD), and the percentage of normal RR intervals that differ by 50 ms (pNN50).

OTHER OUTCOMES:
Adverse effects | After 20 minutes of tDCS
  Adverse effects will be evaluated using structured questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Fuad A Hazime, PhD, Principal Investigator — Physical Therapy Department
Locations (1):
- Department of Physical Therapy. Federal University of Piaui, Parnaíba, Piauí, Brazil